CLINICAL TRIAL: NCT05071378
Title: Leveraging Family-Based Assets for Black MSM In House Ball Communities (Our Family, Our Voices-"OFOV)
Brief Title: Leveraging Family-Based Assets for Black MSM In House Ball Communities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: Yale University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Birnbaum MD MPH, Associate Professor of Pediatrics, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1555461; 1R34MH124082-01 (NIH)
Record Dates: First submitted 2021-05-21; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: HIV I Infection
Keywords: Men; House ballroom community; transgender
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: The investigators will determine the feasibility, acceptability and a preliminary estimate of effect size of an evidence-based HIV prevention intervention for Black MSM adapted for HIV status-neutral use with families in the HBC (called: OFOV). The eight-step ADAPT-ITT framework will guide the approach to enhance intervention content to incorporate an asset-building framework. Aim 1 will lead to the combined multi-level intervention adapted to improve congruence with the realities of HBC families. Aim 2 will assess the feasibility and acceptability of conducting a cluster randomized controlled trial of OFOV with a standard of care wait-listed control group. Data collected from the CRCT will be used to estimate the effect size of OFOV on HIV testing and PrEP use (primary outcome for HIV-negative participants), HIV care engagement and use of ARV treatment (primary outcome for PLHIV), as well as number of family-based assets and sexual health measures (status-neutral secondary outcomes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): This arm will be enrolled in the intervention prior to any data collection
  Interventions: Behavioral: Our Family, Our Voices
- Wait listed control (No Intervention): This arm will receive the intervention after all study data is collected

INTERVENTIONS:
Behavioral: Our Family, Our Voices — Many Men, Many Voices (3MV) is a seven-session, group-level intervention developed to prevent HIV and sexually transmitted diseases (STDs) among black men who have sex with men (MSM) who may or may not identify themselves as gay. The intervention addresses factors that influence the behavior of black MSM: cultural, social, and religious norms; interactions between HIV and other STDs; sexual relationship dynamics; and the social influences that racism and homophobia have on HIV risk behaviors. Our Family, Our Voices seeks to create an adaptation of Many Men, Many Voices specifically tailored to young people who are members of the house ball community by incorporating elements of family support and resilience afforded to participants in the intervention.
  Other Names: an adaptation of Many Men, Many Voices
  Arms: Intervention Group

SUMMARY:
Despite the advent of highly effective prevention tools such as HIV pre-exposure prophylaxis (PrEP), Black men who have sex with men (MSM) continue to have the highest incidence of new HIV diagnoses in the US but are least likely to be engaged in care or to be virally suppressed. Many Black MSM face multiple stigmas but some have found refuge in the House Ball Community (HBC)-a national network of Black LGBT kinship commitments (families) that provide (informal) care giving, affirmation and survival skills-building for its members. The HBC is a large, yet underserved, community within the larger LGBT community. The investigators propose to modify a well-established skills-building and HIV prevention best-evidence, group-level intervention for HIV-negative Black MSM, Many Men Many Voices, into a family-based intervention to focus on asset-building for both HIV-negative and HIV-positive Black MSM within HBC families. Many Men Many Voices (3MV) is a six-session, group-level behavioral intervention and is the only "best evidence" intervention for Black MSM. Family-based interventions have shown HIV prevention efficacy; however, 3MV is not a family-based intervention. In 3MV, HIV-negative Black MSM are recruited into artificial group settings with individuals with whom they may have little social relationship. 3MV neither leverages the connections and commitments nor addresses the variability in HIV-status that exists in house ball families. Because Black MSM in the HBC have closer social relationships, 3MV requires adaptation to be more responsive to this social structure and dynamic. The study's goal in this clinical trial planning grant is to prepare for a cluster randomized controlled trial (CRCT) to test the effectiveness of the modified 3MV vs. standard of care in reducing new HIV infections and increasing rates of viral suppression among Black MSM in HBC families. The study's central hypothesis is that a modified 3MV intervention incorporating family asset-building will have an amplifying effect on HIV prevention and treatment outcomes. This study will provide necessary data to design and conduct a full-scale CRCT effectiveness trial of OFOV on HIV prevention and care outcomes in Black MSM. By precision-tailoring an evidence-based intervention for the HBC, the investigators' research to improve HIV testing and care engagement will complement national efforts to End the Epidemic by 2030, especially among Black MSM-the highest priority group for domestic HIV prevention.

DETAILED DESCRIPTION:
Although there is access to effective HIV prevention tools such as pre-exposure prophylaxis (PrEP), Black men who have sex with men (MSM) continue to have the highest numbers of new HIV cases in the US and are unlikely to be linked to care or to have their HIV under control. Many Black MSM face many challenges because of racism and homophobia but some have found safety in the House Ball Community -an alternative family network (or houses) for Black LGBT that provide emotional and physical support and care and health information for its members. In this study, the investigators will modify a well-known, six-session group HIV prevention program for HIV-negative Black MSM, called Many Men Many Voices (3MV), and turn it into a family-based program that focuses on Black MSM with and without HIV in House Ball Communities. Family-based group programs have been shown to help prevent individuals from getting HIV; but, 3MV is not a family-based program. And in 3MV, Black MSM without HIV are usually recruited into groups with individuals they have never met before. 3MV doesn't usually use the connections between house ball family members to improve health outcomes and doesn't consider how house ball families have members who are both HIV-negative and HIV-positive. Because Black MSM in the House Ball Community have closer social relationships, 3MV requires modification to better fit the house family structure and how family members interact with each other. The goal in this study is to prepare for a larger study to test if the modified 3MV program works better to reduce new HIV infections and improve the health of HIV-positive Black MSM in the House Ball Community families compared to a no group program.

The investigators predict that a modified version of the 3MV group program for the House Ball Community families will work better than the original version of 3MV on HIV prevention and treatment outcomes. This study will provide important information to help us design and conduct a larger study of this modified version of 3MV called "Our Family Our Voices" on HIV prevention and care outcomes in Black MSM. By tailoring a program for the House Ball Community, this research to improve HIV testing and participation in care will better serve Black MSM-the highest priority group for HIV prevention in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for the study will be determined primarily at the family-level. At least 12 members of the same HBC family must be willing to participate together, of which at least half the participating members must be Black MSM.

Participating family members must reside in the New York City metro area.

Black MSM participants must be at least 18 years old.

Exclusion Criteria:

* Not being a member of a house ballroom community family
* Residing outside the New York City
* Being a member of a house ballroom community family that has been established less than 12 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — At least half of the participating house members must be Black men who have sex with men. Black MSM must also currently self-identify as cisgender or transgender man, report anal sex with another man at least once within the previous six months (note: other HBC family members can identify as any gender).
Enrollment: 168 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
HIV testing | measured at time 0, 3 months and 6 months
  primary outcome for HIV-negative participants: the change in the proportion of those who are HIV-negative having been tested for HIV at the three time point s
HIV testing | measured at time 0, 3 months and 6 months
  primary outcome for HIV-negative participants: total change in the number of HIV test results among those who are HIV-negative and have been tested for HIV at the 3 time points
PrEP use | measured at time 0, 3 months and 6 months
  primary outcome for HIV-negative participants: the change in the proportion of those who are HIV-negative who report taking PrEP at the three time points
HIV care engagement | measured at time 0, 3 months and 6 months
  primary outcome for participants living with HIV: the change in the proportion of those living with HIV who report medical visits at the three time points
Taking ARV treatment | measured at time 0, 3 months and 6 months
  primary outcome for participants living with HIV: the change in the proportion of those living with HIV who report taking ARV treatment at the three time points
Viral load measurement | measured at time 0, 3 months and 6 months
  primary outcome for participants living with HIV: the change in the proportion of those living with HIV with undetectable HIV viral loads among those taking ARV treatment at the 3 time points

SECONDARY OUTCOMES:
Family based assets 1: Sense of Community Scale | measured at time 0, 3 months and 6 months
  The change in the aggregate scores of all study participants across the 3 times points as a secondary measurement to study impact of the intervention
Family based assets 2: READY Tool | measured at time 0, 3 months and 6 months
  The change in the aggregate scores of all study participants across the 3 times points as a secondary measurement to study impact of the intervention
Family based assets 3: Asset Inventory | measured at time 0, 3 months and 6 months
  The change in the Asset Inventory scores of all study participants across the 3 times points as a secondary measurement to study impact of the intervention
Brief Resilience Scale | measured at time 0, 3 months and 6 months
  The change in the aggregate scores of all study participants across the 3 times points as a secondary measurement to study impact of the intervention
Condomless anal intercourse | measured at time 0, 3 months and 6 months
  The change in the relative frequency = # times condoms used during anal sex / total # episodes of anal sex in the past 3 months among all study participants across the 3 times points as a secondary measurement to study impact of the intervention
Number of sexual partners | measured at time 0, 3 months and 6 months
  The change in the total number of sexual partners in the past 3 months among all study participants across the 3 times points as a secondary measurement to study impact of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- HEAT Program/SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No